CLINICAL TRIAL: NCT03833687
Title: Aesthetic Performance and Tolerance Evaluation of an Injective Intradermal Treatment for the Skin Roughness and Laxity of Inner Arm and Abdomen
Brief Title: Aesthetic Performance of an Injective Treatment for the Skin Roughness and Laxity of Inner Arm and Abdomen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Medical Doctor, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E0918
Record Dates: First submitted 2019-02-06; First posted 2019-02-07 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Skin Flaccidity and Roughness of the Abdomen and Inner Arms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Profhilo® (Experimental): The 1st treatment was performed during the basal visit and repeated after 1 month.
  3 mL of Profhilo® for each brachial zone, 1.5 mL for hemiabdomen was injected into the middle-deep dermis by needle (29 G) using a bolus technique called "BAP" (Bio Aesthetic Point technique); this technique involves a series of 10 micro-wheals on 3 horizontal-levels for each tested areas (3-4-3 injection points respectively for the 1st, the 2nd and the 3rd horizontal-level). The amount of product to be injected was of 0.3 ml for each point.
  Interventions: Device: Profhilo®

INTERVENTIONS:
Device: Profhilo® — Profhilo® (IBSA Farmaceutici Italia S.r.l.) is a resorbable medical device 2.25 ml non-pyrogenic pre-filled syringe, containing 2 ml of 3.2% hyaluronic acid for intradermal use (32 mg H-HA + 32 mg L-HA dissolved in 2 ml of saline buffered sodium chloride.

SUMMARY:
The objective of this study was to investigate the aesthetic performance of the Hyaluronic acid (HA)-based dermal filler Profhilo® injected by a novel bio aesthetic point technique ("BAP" technique) in woman aged 40-65 years with mild-moderate skin flaccidity and roughness of the abdomen and inner arms.

ELIGIBILITY:
Inclusion Criteria:

* female sex;
* age 40-65 years;
* 3-4 abdomen and inner arm roughness/laxity grade according to a clinical reference scale;
* asking for abdomen and inner arms laxity and roughness restoration;
* available and able to return to the study site for the post-procedural follow-up examinations;
* accepting to not change their habits regarding food, physical activity, cosmetic and cleansing products for the body;
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes) during the entire duration of the study, without appropriate sun protection;
* accepting to sign the informed consent form.

Exclusion Criteria:

* Pregnancy;
* lactation;
* smokers;
* alcohol or drug abusers;
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study;
* subjects not in menopause who do not accept to perform the pregnancy test at T0 (before the 1st aesthetic procedure) and at T1 (1 month after the 1st injection treatment execution, before the 2nd aesthetic procedure);
* Body Mass Index (BMI) variation (± 1) during the study period;
* performing skin treatments for abdominal and brachial zone aesthetic correction (carboxytherapy injections, body lifting, laser, infrared light, bipolar radiofrequency, vacuum and mechanical massage) in the 6 months prior to the study start;
* aesthetic surgical procedure on abdominal and brachial zone in the past;
* change in the normal habits regarding food, physical activity, cosmetic products and cleansing for the body during the month preceding the test;
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit);
* subjects whose insufficient adhesion to the study protocol is foreseeable;
* participation in a similar study currently or during the previous 6 months.
* Dermatitis;
* presence of cutaneous disease on the tested area, as lesions, scars, malformations;
* recurrent facial/labial herpes;
* clinical and significant skin condition on the test area (e.g. active eczema, psoriasis, severe rosacea, scleroderma, local infections and severe acne).
* Diabetes;
* endocrine disease;
* hepatic disorder;
* renal disorder;
* cardiac disorder;
* pulmonary disease;
* cancer;
* neurological or psychological disease;
* inflammatory/immunosuppressive disease;
* drug allergy.
* Anticoagulants and antiplatelet drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago);
* using of drugs able to influence the test results in the investigator opinion.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline of arm skin roughness and laxity clinical grade | Baseline (T0), 1 month (T1), 4 months (T2)
  Skin roughness and laxity clinical grade, according to a visual score from 1 (no roughness and flaccidity) to 5 (very severe roughness and flaccidity).
Change from baseline of abdomen skin roughness and laxity clinical grade | Baseline (T0), 1 month (T1), 4 months (T2)
  Skin roughness and laxity clinical grade, according to a visual score from 1 (no roughness and flaccidity) to 5 (very severe roughness and flaccidity).
Change from baseline of superficial skin hydration | Baseline (T0), 1 month (T1), 4 months (T2)
  Skin electrical capacitance value was measured mono-laterally on the right or left inner arm and hemiabdomen with Corneometer CM825 (Courage - Khazaka, Köln, Germany). The measure of the skin capacitance properties is an indirect expression of its hydration level.
Change from baseline of deep skin hydration | Baseline (T0), 1 month (T1), 4 months (T2)
  Tissue dielectric constant value of superficial and deep skin layers was measured mono-laterally on the right or left inner arm and hemiabdomen with MoistureMeterD (Delfin Technologies, Kuopio - Finland)
Change from baseline of skin density | Baseline (T0), 1 month (T1), 4 months (T2)
  A little skin area of about 7 cm2 (at level of inner arm was pinched, in standardized conditions, using a specific device. Because of this "pinch" the skin profile changes depending on cutaneous density; when the skin is slack the "pinch" forms a lot of wrinkles. A picture of the skin pinched was taken thanks to Primos compact portable device (GFMesstechnik); Primos software is able to measure skin principal profilometric parameters.
Change from baseline of skin plastoelasticity | Baseline (T0), 1 month (T1), 4 months (T2)
  Superficial and deep skin plastoelasticity was measured mono-laterally on the right or left inner arm and hemiabdomen with the instrument Dermal Torque Meter (Dia-Stron Ltd., UK).
Change from baseline of photographic documentation | Baseline (T0), 1 month (T1), 4 months (T2)
  2D pictures of the abdomen and inner arm

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Milan, MI, Italy